CLINICAL TRIAL: NCT06944535
Title: Efficacy of a Modified Lip Repositioning Surgery Technique With Tie Levator Labii Superioris and Without Frenectomy and Myotomy for Treatment of Excessive Gingival Display: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Other Study IDs: Le Nguyen Lam
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2023-09

CONDITIONS: Excessive Gingival Display
Keywords: Excessive gingival display; gummy smile; ip repositioning surgery
MeSH Terms: interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Modified Lip Repositioning Surgery (Retrospective Cohort): This cohort includes patients who had previously undergone the modified lip repositioning surgery technique without frenectomy and without myotomy. Data were obtained retrospectively from medical records and clinical photographs. No prospective intervention was performed.
  Interventions: Procedure: Modified Lip Repositioning Surgery (Retrospective)

INTERVENTIONS:
Procedure: Modified Lip Repositioning Surgery (Retrospective) — Patients previously underwent a modified lip repositioning surgery technique without frenectomy and without myotomy. For this retrospective study, only existing medical records and clinical photographs were reviewed. No new surgical intervention was performed.

SUMMARY:
This retrospective study aims to evaluate the effectiveness and safety of a modified lip repositioning surgery technique, performed without frenectomy and without myotomy, for the correction of excessive gingival display ("gummy smile"). Data were collected from the medical records and clinical photographs of patients who had previously undergone this surgical procedure at the study site.

DETAILED DESCRIPTION:
Excessive gingival display, commonly referred to as a "gummy smile," is an esthetic concern that may reduce patient satisfaction with their smile and overall facial appearance. Several treatment modalities have been suggested to address this condition, including orthodontic treatment, botulinum toxin injection, and various surgical techniques. Among surgical approaches, lip repositioning surgery has gained popularity due to its minimally invasive nature and ability to provide predictable esthetic outcomes.

A modified lip repositioning technique, performed without frenectomy and without myotomy, has been introduced to reduce morbidity and simplify the procedure while maintaining effectiveness. However, published evidence has largely come from prospective interventional series.

To further evaluate the clinical performance of this modified technique, we conducted a retrospective observational cohort study. Data were obtained from the medical records and clinical photographs of patients who had previously undergone the modified lip repositioning surgery at the study site. No new patients were enrolled and no interventions were prospectively carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with the modified lip repositioning surgery without frenectomy and without myotomy.
* Complete medical records including pre- and post-operative documentation.
* Clinical photographs available before and after surgery.
* Minimum follow-up period documented (≥ 3 months).

Exclusion Criteria:

* The patient has trauma and facial deformities
* Incomplete medical records or missing photographs.
* Patients lost to follow-up before minimum period.
* Patients who had undergone other concurrent surgical/orthodontic procedures affecting gingival display.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had previously undergone modified lip repositioning surgery without frenectomy and without myotomy for the correction of excessive gingival display.
  Data were collected retrospectively from medical records and clinical photographs of eligible patients treated at the study site during the defined study period.
  Only patients with complete documentation before and after surgery were included.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Reduction in gingival display after modified lip repositioning surgery | Baseline and up to 12 months post-surgery
  Measurement of gingival display (in millimeters) on smile, comparing baseline (before surgery) and last available follow-up (after surgery), based on clinical photographs and medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Lam N Le, PhD, Principal Investigator — Can Tho University of Medicine and Pharmacy
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tawfik OK, El-Nahass HE, Shipman P, Looney SW, Cutler CW, Brunner M. Lip repositioning for the treatment of excess gingival display: A systematic review. J Esthet Restor Dent. 2018 Mar;30(2):101-112. doi: 10.1111/jerd.12352. Epub 2017 Nov 27. PMID 29193632